CLINICAL TRIAL: NCT02558387
Title: Phase II Trial of BIBF1120 (Nintedanib) in Patients With Recurrent or Metastatic Salivary Gland Cancer of the Head and Neck : a Multicentre Phase II Study
Brief Title: Trial of BIBF1120 (Nintedanib) in Patients With Recurrent or Metastatic Salivary Gland Cancer of the Head and Neck
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-120133
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Recurrent or Metastatic Salivary Gland Cancer of the Head and Neck
MeSH Terms: conditions — Recurrence | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nintedanib arm (Experimental): Nintedanib has never been applied to salivary gland cancer. Nintedanib was given orally at a dose of 200mg twice daily (bid) until progression or unacceptable toxicity.
  Interventions: Drug: BIBF1120

INTERVENTIONS:
Drug: BIBF1120 — Nintedanib will be given orally at a dose of 200mg twice daily (bid) until progression or unacceptable toxicity.
  Other Names: Nintedanib

SUMMARY:
Recently, sorafenib which can target VEGFR and PDGFR demonstrated 13-16% of response rate in patients with recurrent/metastatic salivary gland cancers, suggesting that VEGFR and PDGFR might be important role in salivary gland cancers. Accordingly, several trials with various anti-angiogenic molecular targeted agents such as dasatinib, dovitinib, or sunitinib in salivary gland cancer are ongoing.

Nintedanib (BIBF1120) is a potent small molecule triple receptor tyrosine kinase inhibitor (PDGFR/ FGFR1-2 and VEGFR1-3). VEGFR-2 is considered to be the crucial receptor involved in initiation of the formation as well as the maintenance of tumor vasculature. In vitro, the target receptors are all inhibited by nintedanib in low nanomolar concentrations. In in vivo nude mouse models, nintedanib showed good anti-tumor efficacy at doses of 50-100mg/kg, leading to a substantial delay of tumor growth or even complete tumor stasis in xenografts of a broad range of differing human tumors.

Based on this background, in this study, the investigators would like to conduct a phase II study of Nintedanib (BIBF 1120) in patients with recurrent or metastatic salivary gland cancer of the head and neck to evaluate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven salivary gland cancer of the head and neck (According to WHO classification, mucoepidermoid cancer, adenoid cystic carcinoma, or adenocarcinoma/salivary duct cancer are eligible)
* Recurrent or metastatic salivary gland cancer of the head and neck patients who failed one line of systemic chemotherapy
* age ≥ 18 years
* At least one measurable tumor lesion according to RECIST 1.1
* ECOG performance status 0-2
* Adequate hematologic function (absolute neutrophil count > 1,500/m/, platelets > 100,000/ml, haemoglobin > 9.0 g/dl), hepatic function (alanine transaminase/aspartate transaminase < 5 x ULN, total bilirubin < 1.5 x ULN), renal function (creatinine clearance > 45 ml/min)
* Written informed consent

Exclusion Criteria:

* Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension, history or myocardial infarction in the 12 months prior to the start of the treatment, or arrhythmia
* Hemorrhagic or thromboembolic events in the past 6 months
* Major injuries in the 10 days prior to start of the study
* Patients with post-obstructive pneumonia or uncontrolled serious infection
* Pregnant or nursing women
* Uncontrolled symptomatic brain metastasis
* Prior history of malignancy within 5 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, and well treated thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
response rate | 6months after patient enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea